CLINICAL TRIAL: NCT01596556
Title: The Effect of Smoking on Thermoregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: International Diabetes Federation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-11-8767-AD-CTIL
Record Dates: First submitted 2012-05-06; First posted 2012-05-11 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Cigarette Smoking
Keywords: smoking; exercise; heat tolerance; heat stroke
MeSH Terms: conditions — Cigarette Smoking; Smoking; Motor Activity; Heat Stroke | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- smokers (Experimental): This arm consists of smokers.
  Interventions: Drug: Nicotine; Other: cigarette smoking
- non-smokers (Active Comparator): non-smoking participants in the study
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — both groups will be given nicotine lozenges before a VO2 test and a HTT.
Other: cigarette smoking — the smokers will smoke 2 cigarettes before a VO2 exam and a HTT.
  Arms: smokers

SUMMARY:
To the best of our knowledge, a possible relation between smoking and heat injuries or heat intolerance was never scientifically examined, although such a relation is logical according to the observations that smoking has a thermogenic effect, decreases physical fitness and affects the body's heat dissipation.16 healthy young male volunteers will participate in the study, 8 smokers and 8 non-smokers. They will arrive to our lab four or six times. They will perform VO2 test and heat tolerance test (HTT) in different conditions.

DETAILED DESCRIPTION:
16 healthy young male volunteers will participate in the study, 8 smokers and 8 non-smokers. They will arrive to our lab four or five times. During their first visit they will go through a VO2 max test in order to evaluate their aerobic fitness, and their physiological efficiency. During their second visit all subjects will go through the same test after exposure to nicotine. During the smokers' third visit they will go through the same test, after exposure to cigarette smoking. During the non-smokers third visit and the smokers fourth visit - they will go through an exercise heat tolerance test without prior smoking. During the fifth visit the smokers will go through an exercise heat tolerance test after exposure to cigarette smoking. During the smokers' sixth visit and the non-smokers fourth visit they will go through an HTT after exposure to nicotine.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* healthy
* after medical checkup
* after signing concent form
* for the smokers: smoking 0.5-1.5 packs of cigarettes a day at least 2 years.

Exclusion Criteria:

* heart disease
* respiratory disease
* baseline bp above 140/90 mmHg
* diabetes
* anhydrosis
* skin disease
* acute illness
* detoxification from nicotine
* allergy to nicotine
* smoking other then specified in the inclusion criteria

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Heat tolerance | 2-3 days
  The test is performed in a climatic chamber at a temperature of 40oC and 40% relative humidity. During the test, the subject walks on a treadmill at a speed of 5 km/hr at a 2% grade for 2h. Body core temperature and heart rate are continuously monitored, and sweat rate is computed from body weight prior to and after the test, corrected for fluid intake. Heat intolerance is determined when body core temperature elevates above 38.5oC, when heart rate elevates above 150 bpm, or when either does not tend to reach a plateau.
VO2max | 2-3 days
  volunteer's oxygen consumption (VO2) will be monitored continuously with a metabolic chart (ZAN), while running for 10 min on a treadmill under comfortable environmental conditions.

SECONDARY OUTCOMES:
Rectal temperature | experimental days 4,5,6
  The volunteers will undergo heat tolerance test. Their rectal temperature will be measured by rectal thermistor and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system
Heart rate | experimental days 4,5,6
  During the HTT and the VO2 test heart rates will be monitored continuously and will be stored by a heart rate wristwatch, (POLAR, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Druyan, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- The Institute of Military Physiology Heller Institute of Medical Research, Tel-Hashomer Ramat-Gan, Israel